CLINICAL TRIAL: NCT01119391
Title: The Impact of Lifestyle Behaviors on IVF Outcome
Brief Title: The Impact of Lifestyle Behaviors on In Vitro Fertilization (IVF) Outcome
Status: Completed | Type: Observational
Sponsor: Boston IVF (Other)
Responsible Party: Principal Investigator, Alice D. Domar, PhD, Alice D. Domar, PhD, Boston IVF
Other Study IDs: 20091005
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: IVF; Lifestyle habits
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing IVF: Women undergoing an in vitro fertilization cycle
  Interventions: Behavioral: There was no intervention; this was a survey only study

INTERVENTIONS:
Behavioral: There was no intervention; this was a survey only study — There was no intervention; this was a survey only study

SUMMARY:
Many women undergoing in vitro fertilization (IVF) ask their doctor if there are any behaviors they should avoid, or any behaviors they should emphasize during their IVF cycle. This study examines the effects of health habits surrounding exercise, smoking, alcohol, sleep, caffeine, herbal medications, acupuncture, and diet on pregnancy rates during IVF cycles. The purpose of this study is to determine if lifestyle behaviors have a significant impact on pregnancy rates during treatment with IVF.

This is an observational study conducted at a private academically-affiliated infertility clinic and includes 118 women ages 44 and below scheduled to undergo IVF treatment. All subjects were asked to complete a health history survey at the time of enrollment and a daily survey during each day of their IVF cycle. The primary outcome is clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Female Boston IVF infertility patient undergoing IVF treatment
* Age 18-44 years
* Able to read, understand and sign the informed consent in English
* Willing and able to comply with study requirements
* Must be well versed in using a personal computer and the internet and must have access to an internet-connected computer seven days per week

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women about to undergo an in vitro fertilization cycle at Boston IVF
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rates | Approximately 28 days (1 IVF cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Alice D Domar, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domar AD, Conboy L, Denardo-Roney J, Rooney KL. Lifestyle behaviors in women undergoing in vitro fertilization: a prospective study. Fertil Steril. 2012 Mar;97(3):697-701.e1. doi: 10.1016/j.fertnstert.2011.12.012. Epub 2012 Jan 3. PMID 22217965